CLINICAL TRIAL: NCT07179523
Title: Randomized Clinical Evaluation of the Effectiveness of Biomimetic Hemostatic Sponges ColiSorB Following Dental Extraction
Brief Title: Clinical Evaluation of the Effectiveness of Biomimetic Hemostatic Sponges ColiSorB Following Dental Extraction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sara Omar (Other)
Collaborators: Incura Inc. (Other)
Responsible Party: Sponsor-Investigator, Sara Omar, Clinical Researcher, The American University in Cairo
Organization: The American University in Cairo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26522
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Molar Extraction Socket
Keywords: ColiSorB
MeSH Terms: interventions — Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Conventional cotton and gauze were applied with firm pressure on the extraction site
- Experimental Comparator Group (Active Comparator): A commercially available hemostatic sponge was used, namely Cutanplast.
  Interventions: Combination Product: Hemostatic Agent
- Experimental Group (Experimental): A newly developed hemostatic gelatin sponge called Colisorb was used
  Interventions: Combination Product: Hemostatic gelatin sponge

INTERVENTIONS:
Combination Product: Hemostatic gelatin sponge — Colisorb® exhibits optimal pore structure, number and size, which results in its structure being highly porous with low density. In addition, Colisorb® possesses optimal mechanical integrity allowing it to swell to its maximal absorption capacity while maintaining mechanical stability. The sponge can absorb fluids in the blood resulting in prompt recruitment of clotting factors, hence accelerating the body's natural blood clotting cascade. Colisorb® was configured in a way to imitate natural adhesive mechanism without the use of co-agulants, it provides a safer and a more efficient alternative for minimizing post-operative complications and enhancing recovery. Upon performing the tooth extraction, oral surgeon instantly applied the sponge. Patients were prescribed, antibiotics, and antacid, if needed, for 3 days and analgesics for 5 days, followed by a mouth wash routine of warm water with salt to enhance healing outcomes. Patients visited the clinic three days after surgery.
  Arms: Experimental Group
Combination Product: Hemostatic Agent — Gelatin sponge that may be soaked with sterile physiological solution. Biocompatible and easy to use for 5 to 10 minute bleeding control rate.
  Upon performing the tooth extraction, oral surgeon instantly applied the sponge in the socket where the tooth was extracted to facilitate hemostasis. Patients were prescribed, antibiotics, and antacid, if needed, for 3 days and analgesics for 5 days, followed by a mouth wash routine of warm water with salt to enhance healing outcomes. Patients visited the clinic three days after surgery.
  Other Names: Cutanplast
  Arms: Experimental Comparator Group

SUMMARY:
This study tested three different treatment groups in a fair and organized way. It included people who came to Cairo University's Dental Department to have a back tooth (molar) removed and who qualified to join.

Out of 40 people who were checked, 8 did not meet the requirements, and 2 others did not return for check-up visits.

The study followed all ethical rules and was approved by the Research Ethics Committee at Cairo University's Faculty of Oral and Dental Medicine.

DETAILED DESCRIPTION:
ColiSorB® is a novel biomimetic adhesive, coagulant-free hemostatic sponge engineered for dental and surgical applications. Unlike conventional hemostatic methods that rely on mechanical compression or exogenous coagulation agents, ColiSorB® mimics the body's natural adhesive and clot-stabilization mechanisms. Its architecture replicates the fibrin mesh, forming a bio-adhesive matrix at the application site to achieve rapid hemostasis, minimize patient discomfort, and reduce postoperative complications such as persistent bleeding and alveolar osteitis (dry socket).

The material is composed of a gelatin-based, non-pyrogenic, absorbable polysaccharide that is both cost-effective and adaptable. By eliminating the need for coagulants, ColiSorB® offers a simplified, biocompatible approach to bleeding control in dental extractions.

This study aimed to evaluate the safety and effectiveness of ColiSorB® sponges in patients undergoing molar extraction, with direct comparison to both a widely used commercial reference product (Cutanplast®) and the conventional method of gauze or cotton under pressure. The primary endpoint was the achievement of post-extraction hemostasis, while secondary endpoints included assessment of postoperative pain and wound healing.

Study Groups

Participants were randomized into three equal groups (n = 10 per arm):

1. Test group: ColiSorB® hemostatic sponge.
2. Comparator group: Cutanplast®, a commercially available gelatin-based hemostatic product.
3. Control group: Conventional method using sterile gauze under biting pressure.

A total of 30 extraction sites were evaluated, with each group receiving its designated hemostatic intervention immediately following extraction.

Application and Assessments

* Hemostatic efficacy: Time to complete hemostasis was recorded, with success rates measured at 3 and 10 minutes.
* Bleeding assessment: Bleeding severity was scored using a visual analogue scale (VAS).
* Safety outcomes: Postoperative complications (e.g., infection, dry socket, persistent bleeding), periodontal integrity, and radiographic findings were monitored on postoperative days 1 and 7.
* Pain outcomes: Postoperative pain was evaluated using VAS scores at days 1 and 7.

The study protocol was approved by the Research Ethics Committee, and informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria

* Patients seeking removal of a wisdom tooth due to:
* Severe decay
* Malposition/misalignment
* Pressure caries affecting adjacent teeth
* Indication for future orthodontic treatment
* Age ≥ 14 years
* Available for at least one postoperative evaluation (scheduled approximately 7 days post-surgery)
* Willing and able to provide informed consent for participation

Exclusion Criteria

* Unwillingness to provide informed consent
* Current use of anticoagulant medications (e.g., Aspirin, Coumadin, Plavix) or discontinuation of such medications < 3 days prior to surgery
* Pregnant, planning pregnancy during the follow-up period, or actively breastfeeding
* Active or suspected infection at the surgical site
* Known sensitivity or allergy to any component of the hemostatic gelatin sponge
* Severe congenital or acquired immunodeficiency
* Undergoing bisphosphonate therapy
* Diabetes with unstable blood glucose levels

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Time to achieve full absorption and hemostasis | Assessed from baseline until hemostasis is achieved (within 1 day).
  Time (in minutes) from baseline (application of the assigned dressing immediately after tooth extraction) until complete hemostasis is achieved, defined as cessation of visible bleeding at the extraction site.
Time of placement | Assessed at baseline (time of dressing application immediately after tooth extraction).
  Duration (in minutes) required at baseline to apply the assigned dressing (sponge or standard gauze) at the extraction site, including any pre-wetting step if applicable.

SECONDARY OUTCOMES:
Pain and Healing Scale | Up to 7 days
  Patients comfort level is assessed by a verbal inquiry after completion of the operation and dressing application ( post- operation).
  Pain scores: Patient-reported pain scores assessed on day 1, and day 7 of post-procedure appointment. Based on a 0 to 10 self-reported pain score basis, with 0 being no pain and 10 being the worst pain the patient had ever experienced.
  Healing: Sealing of the wound was assessed on day 1, and day 7 post-operation. Using a modified scale adopted from Landry, Turnbull and Howley healing Index. The parameters based on which the wound sealing is assessed include tissue color, bleeding on palpation, granulation tissue, incision margin and suppuration. The adjusted scale was as follows: 1 (significantly getting worse or very poor), 2 (moderate), and 3 (significantly better or excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral & maxillofacial surgery at Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study. The data are considered the property of the study sponsor and the collaborator, will remain confidential.